CLINICAL TRIAL: NCT05462275
Title: Impact of Patient Position on the Success in Placing Triple-cuffed Double Lumen Endotracheal Tube : Multi-center Observational Study
Brief Title: Impact of Patient Position on the Success in Placing Triple-cuffed Double Lumen Endotracheal Tube
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hansu Bae (Other)
Responsible Party: Sponsor-Investigator, Hansu Bae, Assistant professor, Dongguk University International Hospital
Organization: Dongguk University International Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Ankor-1
Record Dates: First submitted 2022-07-06; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Lung Diseases
Keywords: 3-cuffed double lumen tube; one lung ventilation; lung isolation
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: Interventional observational study. The investigators conduct this study to analyze the impact of patient position on the success in placing triple-cuffed double lumen endotracheal tube.
Masking Description: This study don't require any types of masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental): There is only one group to evaluate this observational study.
  Interventions: Device: Intubation using 3-cuffed double lumen endotracheal tube

INTERVENTIONS:
Device: Intubation using 3-cuffed double lumen endotracheal tube — After patient's position, 3-cuffed double lumen endotracheal tube is intubated without fiberoptic bronchoscopy guidance

SUMMARY:
Triple-cuffed double lumen endotracheal tube (TC-DLT, ANKOR tube. Insung corp., Korea) which was developed to isolate lung without endotracheal bronchoscope guidance has additional carinal cuff placed between bronchial tube cuff and tracheal tube cuff. This device has been successfully used to isolate lung more simply in specific settings when there is too much excretion to visualize endotracheal structure or for a health provider who is not good at use of traditional double-lumen tube. Although TC-DLT is designed to enable lung separation effectively in situations that confirmation of tube position using bronchoscopy is difficult or not available, but no studies have been conducted on whether effective lung isolation using TC-DLT is possible after change in the relative position of the bronchial tree by postural change. This plan was prepared for research on this.

DETAILED DESCRIPTION:
After enter into operating room, induction of anesthesia is performed through standard general anesthesia procedure before endotracheal intubation. Endotracheal intubation is performed using TC-DLT and inflate carinal cuff with 5 ~ 15ml of air. Then, push it into trachea until resistance is felt. When carinal cuff is placed at carina, deflate carinal cuff and isolate independent lung followed by confirmation of bronchial cuff position using fiberoptic bronchoscopy.

Record the location of the bronchial balloon in one of the following conditions

1. at proper position(proximal upper end of bronchial balloon is between 5mm from carinal opening) :
2. proximal end of bronchial balloon is placed more of 5mm distally from carinal opening
3. proximal end of bronchial balloon is placed more of 5mm proximally from carinal opening

Then, change patient position to left lateral decubitus (LLD) position and check the position of bronchial balloon using fiberoptic bronchoscopy as previously done.

1. at proper position(proximal upper end of bronchial balloon is between 5mm from carinal opening) :
2. proximal end of bronchial balloon is placed more of 5mm distally from carinal opening
3. proximal end of bronchial balloon is placed more of 5mm proximally from carinal opening

After check whether there is something to considerate, end this case.

ELIGIBILITY:
Inclusion Criteria:

* Adults who is including in ASA class I or II
* Patients scheduled for right lung surgery under right lung isolation
* Patients who don't have any anatomical variations in pulmonary system
* Patients who have never gotten a lung surgery

Exclusion Criteria:

* Pregnancy
* Patients who are predicted difficult intubation
* Patients who is under upper airway infection
* Patients who have coagulopathy
* Emergency surgery
* In addition, patients considered inappropriate to participate in this study

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-04-29 (Estimated); Study Completion 2023-04-29 (Estimated)

PRIMARY OUTCOMES:
Success rate of 3-cuffed double lumen tube inserted in lateral position | During procedure(Immediately after secondary intubation)
  Authors insert 3-cuffed double lumen tube after position change to left lateral decubitus with blind fashion. At this time, probability that the tube will be inserted to an appropriate depth is primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Dongkyu Lee, Study Chair — Department of anesthesiology, Dongguk University Il-san hospital
Locations (1):
- Dongguk University Il-san hospital, Goyang-si, Geyonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
This study is multi center observational study and we will not share any patients data with other center

REFERENCES:
- [Background] Boisen ML, Schisler T, Kolarczyk L, Melnyk V, Rolleri N, Bottiger B, Klinger R, Teeter E, Rao VK, Gelzinis TA. The Year in Thoracic Anesthesia: Selected Highlights from 2019. J Cardiothorac Vasc Anesth. 2020 Jul;34(7):1733-1744. doi: 10.1053/j.jvca.2020.03.016. Epub 2020 Apr 18. PMID 32430201
- [Background] Boisen ML, Fernando RJ, Kolarczyk L, Teeter E, Schisler T, La Colla L, Melnyk V, Robles C, Rao VK, Gelzinis TA. The Year in Thoracic Anesthesia: Selected Highlights From 2020. J Cardiothorac Vasc Anesth. 2021 Oct;35(10):2855-2868. doi: 10.1053/j.jvca.2021.04.012. Epub 2021 Apr 17. PMID 34053812
- [Background] Seo Y, Kim N, Paik HC, Park D, Oh YJ. Successful blind lung isolation with the use of a novel double-lumen endobronchial tube in a patient undergoing lung transplantation with massive pulmonary secretion: A case report. Medicine (Baltimore). 2019 Aug;98(33):e16869. doi: 10.1097/MD.0000000000016869. PMID 31415423
- [Background] Kim N, Byon HJ, Kim GE, Park C, Joe YE, Suh SM, Oh YJ. A Randomized Controlled Trial Comparing Novel Triple-Cuffed Double-Lumen Endobronchial Tubes with Conventional Double-Lumen Endobronchial Tubes for Lung Isolation. J Clin Med. 2020 Apr 1;9(4):977. doi: 10.3390/jcm9040977. PMID 32244659
- [Background] Ball WS, Wicks JD, Mettler FA Jr. Prone-supine change in organ position: CT demonstration. AJR Am J Roentgenol. 1980 Oct;135(4):815-20. doi: 10.2214/ajr.135.4.815. PMID 6778119